CLINICAL TRIAL: NCT01059500
Title: Quantitative Pretest Probability to Reduce Cardiopulmonary Imaging in the ED
Brief Title: Assessment of Acute Disease to Reduce Imaging Costs
Acronym: QUAADRICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R18HS018519-01 (AHRQ)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-11

CONDITIONS: Acute Coronary Syndrome; Pulmonary Embolism
Keywords: Computer-derived, quantitative pretest probability (PTP); Overtesting; Radiation; Intravenous Contrast; Anticoagulation
MeSH Terms: conditions — Acute Coronary Syndrome; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Webtool Output (Experimental): The webtool output group will receive the numeric PTP estimate from webtool output.
  Interventions: Device: Webtool
- Standard of Care/No Webtool Output (No Intervention): The control group will not receive the numeric PTP estimate.

INTERVENTIONS:
Device: Webtool — Webtool provides the numeric PTP estimate for ACS and PE, and one of three testing recommendations. For ACS, PTP <2.5% with low clinical suspicion and available follow-up, no further testing; PTP 2.5 to 5.5%: obtain a troponin I measurement at presentation and 120 minutes later, and if both are normal, no further testing; PTP >5.5%: proceed to provocative testing. For PE, PTP<2.5% with low clinical suspicion and available follow-up, no further testing; PTP 2.5-10%, obtain a quantitative D-dimer and if normal, no further testing. PTP 10-20%, proceed directly to pulmonary vascular imaging, and if PTP>20% consider empiric anticoagulation with heparin if no contraindications.
  Arms: Webtool Output

SUMMARY:
Overtesting for Acute Coronary Syndrome(ACS) and Pulmonary Embolism (PE) in low risk Emergency Department(ED) patients can increase exposure of nondiseased patients to radiation, intravenous contrast and anticoagulation. This project addresses question of whether quantitative Pre-Test Probability(PTP) assessed from two validated web-based computer algorithms (the project "webtool"), can improve the diagnostic evaluation of adult patients with charted evidence of chest pain and dyspnea. After a validation phase, the main study will randomize patients to either the Standard care group or the Intervention group, which will receive the output of the ACS and PE webtool that includes the PTP estimates of ACS and PE and one of three recommendations regarding next steps: 1. No further testing, 2. Exclusion with a biomarker protocol, or 3. Immediate imaging +/- empiric anticoagulation.

ELIGIBILITY:
Inclusion Criteria

* Adult (>17 years) ED patient reports a history of chest discomfort and new or worsened shortness of breath or breathing difficulty, documented in the written history of present illness or review of systems.
* Patient must understand English or have a certified translator present.
* Physician has ordered or plans to order a 12-lead electrocardiogram.
* Patient indicates the site hospital was his or her "hospital of choice" in the event of return visit within 14 days.

Randomization Exclusions

* Positive urine cocaine test.
* Incarceration within 14 days of enrollment.
* Patient elopement from medical care (i.e., patients who leave against medical advice).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Kline, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Carolinas Medical Center, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peitz GW, Troyer J, Jones AE, Shapiro NI, Nelson RD, Hernandez J, Kline JA. Association of body mass index with increased cost of care and length of stay for emergency department patients with chest pain and dyspnea. Circ Cardiovasc Qual Outcomes. 2014 Mar;7(2):292-8. doi: 10.1161/CIRCOUTCOMES.113.000702. Epub 2014 Mar 4. PMID 24594550
- [Derived] Kline JA, Jones AE, Shapiro NI, Hernandez J, Hogg MM, Troyer J, Nelson RD. Multicenter, randomized trial of quantitative pretest probability to reduce unnecessary medical radiation exposure in emergency department patients with chest pain and dyspnea. Circ Cardiovasc Imaging. 2014 Jan;7(1):66-73. doi: 10.1161/CIRCIMAGING.113.001080. Epub 2013 Nov 25. PMID 24275953
- [Derived] Kline JA, Shapiro NI, Jones AE, Hernandez J, Hogg MM, Troyer J, Nelson RD. Outcomes and radiation exposure of emergency department patients with chest pain and shortness of breath and ultralow pretest probability: a multicenter study. Ann Emerg Med. 2014 Mar;63(3):281-8. doi: 10.1016/j.annemergmed.2013.09.009. Epub 2013 Oct 10. PMID 24120629
- [Derived] Kline JA, Stubblefield WB. Clinician gestalt estimate of pretest probability for acute coronary syndrome and pulmonary embolism in patients with chest pain and dyspnea. Ann Emerg Med. 2014 Mar;63(3):275-80. doi: 10.1016/j.annemergmed.2013.08.023. Epub 2013 Sep 23. PMID 24070658
- See also: Article "Multicenter, randomized trial of quantitative pretest probability to reduce unnecessary medical radiation exposure in emergency department patients with chest pain and dyspnea" — https://pubmed.ncbi.nlm.nih.gov/24275953/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 550 subjects signed consent. 8 subjects screenfailed. 1 subject withdrew consent. 541 subjects were randomized.
Period: Overall Study
Arm/Group | Webtool Output | Standard of Care/No Webtool Output
Started | 264 | 277
Completed | 264 | 277
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Webtool Output | Standard of Care/No Webtool Output | Total
Number analyzed (Participants) | 264 | 277 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15) | 49 (14) | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 149 | 303
  Male | 110 | 128 | 238
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 124 | 148 | 272
  Unkown or Not reported | 140 | 129 | 269
Region of Enrollment [Number; unit: participants]
  United States | 264 | 277 | 541

OUTCOME MEASURES:

1. Primary Outcome: Efficiency--Mean Cost of Care
Description: Only costs at the enrollment hospital will be used, and only for patients who indicate that they did not visit any other hospital at the time of phone follow-up. Costs would exclude unexpected and unrelated events such as trauma. Additionally, estimated costs associated with the time required of the clinician to gather and enter the 17 variables are included.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Standard of Care/No Webtool Output | Webtool Output
Number analyzed (Participants) | 277 | 264
US Dollars | 3933 (12639) | 2761 (7965)

2. Secondary Outcome: Efficiency--Total Charge of Medical Care
Description: Amount charged for medical care.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Standard of Care/No Webtool Output | Webtool Output
Number analyzed (Participants) | 277 | 264
US Dollars | 16413 (38993) | 11916 (26288)

3. Secondary Outcome: Safety--Radiation Dose to the Chest
Description: in millisievert (mSv)
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: mSv
Arm/Group | Standard of Care/No Webtool Output | Webtool Output
Number analyzed (Participants) | 277 | 264
mSv | 5.2 (7.0) | 4.2 (6.0)

4. Secondary Outcome: Effectiveness--Length of Stay in Hospital
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard of Care/No Webtool Output | Webtool Output
Number analyzed (Participants) | 277 | 264
hours | 31.7 (63.3) | 27.1 (74.6)

5. Secondary Outcome: Effectiveness--Length of Stay Emergency Department
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Standard of Care/No Webtool Output | Webtool Output
Number analyzed (Participants) | 277 | 264
Hours | 5.7 (2.5) | 5.7 (3.0)

ADVERSE EVENTS:
Time Frame: Baseline through Day 90
Arm/Group | Webtool Output | Standard of Care/No Webtool Output
All-Cause Mortality (participants affected / at risk) | 0/264 | 2/277
Serious Adverse Events (participants affected / at risk) | 34/264 | 49/277
Other Adverse Events (participants affected / at risk) | 0/264 | 0/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Webtool Output (N=264) | Standard of Care/No Webtool Output (N=277)
death (General disorders) | 0 (0) | 1 (1)
death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 2 (2) | 4 (4)
syncope (General disorders) | 1 (1) | 1 (1)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
anemia (Vascular disorders) | 1 (1) | 1 (1)
bile leak (Hepatobiliary disorders) | 1 (1) | 0 (0)
non-ST-elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 5 (5) | 4 (4)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
acute worsening of abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
left sided neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
congestive heart failure (Cardiac disorders) | 2 (2) | 0 (0)
restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
pulmonary embolism (Vascular disorders) | 2 (2) | 7 (7)
gastric ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
worsening abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
right rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
right bicep repair (Surgical and medical procedures) | 1 (1) | 0 (0)
tenosynovitis repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Group B streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 1 (1) | 1 (1)
cocaine induced chest pain (Cardiac disorders) | 1 (1) | 0 (0)
cocaine induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
bronchiectasis pseudomas pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
unstable angina (Cardiac disorders) | 1 (1) | 1 (1)
acute alcohol withdrawal (General disorders) | 1 (1) | 0 (0)
alcohol dependence (General disorders) | 1 (1) | 0 (0)
mixed state bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
noncompliance with medical treatment (General disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
non-small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
bone pain from lytic lesions secondary to multiple myeloma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dermatomyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
metastatic adenocarcinoma of the left humerus causing pathological fracture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
liver hematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
coronary artery bypass grafting (Cardiac disorders) | 1 (1) | 0 (0)
left ventricular thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
ST-elevation myocardial infarction (STEMI) (Cardiac disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
lower extremity bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
multiple myeloma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hypertensive urgency (Cardiac disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 0 (0) | 2 (2)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
planned elective electrophysiology study (Surgical and medical procedures) | 0 (0) | 1 (1)
atrial flutter ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
gall stone pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
hospitalization for unknown reason (General disorders) | 0 (0) | 1 (1)
severe vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
severe diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
congestive heart failure exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
lymphocytic leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
skin fungal infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
right femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lupus flare (Immune system disorders) | 0 (0) | 1 (1)
vitamin D deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
iron deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
spina bifida occulta (Nervous system disorders) | 0 (0) | 1 (1)
post right popliteal superficial femoral thrombectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
accute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
malignant polyp within the sigmoid colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
atypical chest pain (Cardiac disorders) | 0 (0) | 1 (1)
intentional drug overdose (Psychiatric disorders) | 0 (0) | 2 (2)
dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
benign right lobe lung nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
lower extremity paralysis (Nervous system disorders) | 0 (0) | 1 (1)
diuresis (Renal and urinary disorders) | 0 (0) | 1 (1)
heart catheterization (Surgical and medical procedures) | 0 (0) | 2 (2)
heart failure (Cardiac disorders) | 0 (0) | 1 (1)
esophagogastrodeudenoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
deep vein thrombosis in right lower extremity and right common femoral vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No